CLINICAL TRIAL: NCT02972970
Title: Feasibility Study to Assess the Scan, Fit and Print Process for the Aveera "Patient Matched" CPAP Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metamason (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Meta-001
Record Dates: First submitted 2016-11-09; First posted 2016-11-25 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aveera (Other): This is a prospective, open label study to assess the scan, print and fit process to see if the Aveera will be able to be used with conventional CPAP therapy devices
  Interventions: Device: Aveera

INTERVENTIONS:
Device: Aveera — Subjects will use the 3D crafted CPAP mask. All subjects will receive a mask to use

SUMMARY:
Feasibility study to assess the scan, fit and print process for the Aveera "Patient Matched" CPAP Mask

DETAILED DESCRIPTION:
1. Assess the process of scan, fit and print
2. Subjective/objective assessment of fit of the Aveera during the 2 week use for leaks and comfort
3. Ethnographic insights into the user experience of the scan, fit, print process.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Both genders
* Currently prescribed fixed pressure CPAP or APAP for the treatment of OSA
* Currently CPAP pillows and nasal mask users
* Patients who are adherent as defined by conventional standards (i.e. 4 hours per night/70% of the nights)

Exclusion Criteria:

* Unwilling to wear the AVEERA
* Concern about privacy of data
* Pregnant
* Full face mask user
* Any medical condition deemed by the investigator to pose an issue with the subject's participation.
* Upper limit of CPAP pressure of ≥ to 15 cm H20 or APAP a upper limit pressure setting of ≥17cm H2O
* Requires the use of supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
1) Measure time frame from scanning to mask fit and subjective patient feedback of mask fit | 2 weeks
  Assess the clinical utility of using a 3D scanning process, printing and fit assessment

CONTACTS AND LOCATIONS:
Overall Officials: robyn woidtke, Study Director — Consultant
Locations (1):
- Tower Sleep Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual data